CLINICAL TRIAL: NCT01527500
Title: A Multicenter, Randomized, Sham-control, Proof-of-concept Study of Intravitreal LFG316 in Patients With Geographic Atrophy Associated With Age-related Macular Degeneration
Brief Title: Intravitreal LFG316 in Patients With Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLFG316A2203
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Geographic Atrophy; Age-related Macular Degeneration
Keywords: AMD; Age-related Macular Degeneration; geographic atrophy; GA; Dry AMD; Blindness; Drusen; GA lesion
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration; Blindness | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- LFG316 higher dose (Experimental): LFG316 10 mg/100 μL
  Interventions: Drug: LFG316
- Sham (Sham Comparator): Sham injection
  Interventions: Drug: Sham
- LFG316 lower dose (Experimental): LFG316 5 mg/ 50 μL
  Interventions: Drug: LFG316 Lower dose

INTERVENTIONS:
Drug: LFG316 — LFG316 5 mg/50 μL solution for IVT injection,
  Arms: LFG316 higher dose
Drug: Sham — Sham injection (akin to intravitreal injection but without intravitreal needle; no investigational drug given)
  Arms: Sham
Drug: LFG316 Lower dose — LFG316 5 mg/50 μL solution for IVT Injection
  Arms: LFG316 lower dose

SUMMARY:
This study was conducted in two parts; Part A and Part B: Part B was initially planned to include two cohorts. Cohort 2 was cancelled following an interim analysis for efficacy in Part A of the study, and not due to any safety issues or concerns. Cohort 2 is not referred to again and part B cohort 1 is referred to as part B alone in the remainder of the document and is the subject of this report.

Part B was conducted to assess the safety and tolerability of a single intravitreal (IVT) LFG316 10 mg/100 µL injection. There was no efficacy evaluation in Part B. The study employed a multicenter, randomized, sham - controlled, single masked design. Eight patients with advanced AMD were planned to be randomized in a 3:1 ratio to receive a single IVT dose of LFG316 (10 mg/100 µL) or sham injection. Patients assigned to a sham injection were treated the same as those assigned to LFG316, except that the hub of an empty syringe (without needle) was placed against the eye instead of the IVT injection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AMD if enrolled in Part B of study
* Geographic atrophy in at least one eye if enrolled in Part A of study
* ETDRS best corrected visual acuity of 60 letters or worse (~≤ 20/63)

Exclusion Criteria:

* Retinal disease other than AMD
* History of choroidal neovascularization
* Severe cataract
* History of infectious uveitis or endophthalmitis
* Eye surgery in the non-study eye within 30 days prior to study
* Eye surgery or IVT injection in the study eye within 90 days prior to study
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-01-25 (Actual); Primary Completion 2015-06-24 (Actual); Study Completion 2015-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (18):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Winter Haven, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Leawood, Kansas
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Grand Rapids, Michigan
  - Novartis Investigative Site, Jackson, Michigan
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Silverdale, Washington

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted in 2 parts: Part A & Part B.
  Part A evaluated safety & efficacy of multiple 5 mg/50 µL doses of intravitreal (IVT) LFG316 against sham every 28 days for 505 days
  Part B evaluated the safety and pharmacokinetics of a single IVT dose of 10 mg/100 µL of LFG316
Period: Part A
Arm/Group | LFG316 | Sham
Started | 99 | 51
Completed | 69 | 38
Not Completed | 30 | 13
Not completed — Administrative | 11 | 7
Not completed — Adverse Event | 4 | 2
Not completed — Death | 4 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Deviation | 9 | 2
Not completed — Withdrawal by Subject | 2 | 0
Period: Part B
Arm/Group | LFG316 | Sham
Started | 7 | 1
Completed | 6 | 1
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A- LFG316 5 mg: LFG316 5 mg injection every 28 days for a total of 12 injections
- Part A- Sham: sham injection every 28 days for a total of 12 injections
- Part B- LFG316 10 mg: Single LFG316 10 mg Injection
- Part B- Sham: Single Sham injection
- Total: Total of all reporting groups
Arm/Group | Part A- LFG316 5 mg | Part A- Sham | Part B- LFG316 10 mg | Part B- Sham | Total
Number analyzed (Participants) | 99 | 51 | 7 | 1 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] — PART A (N=99, 51), LFG316 (5 mg/50 µL), sham injection every 28 days for 505 days. PART B (N=7, 1), LFG316 (10 mg/100 µL), single sham injection
  years | 78.6 (7.5) | 80.8 (6.5) | 84.1 (3.8) | 81.0 (NA) — Only a single participant was analyzed therefore there is no SD (NA) | 79.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants] — PART A (N=99, 51), LFG316 (50 mg/50 µL), sham injection every 28 days for 505 days. PART B (N=7, 1), LFG316 (10 mg/100 µL), single sham injection
  Participants
    Female | 58 | 32 | 6 | 1 | 97
    Male | 41 | 19 | 1 | 0 | 61

OUTCOME MEASURES:

1. Primary Outcome: Part A: Geographic Atrophy (GA) Lesion Growth Measured by Fundus Autofluorescence (FAF) From Baseline to Day 505
Description: Geographic atrophy (GA) lesion growth measured by fundus autofluorescence (FAF) from baseline to Day 505.
Time Frame: Day 1 to Day 505 (starting from the day of first intravitreal injection until Day 505)
Population: Pharmacodynamic analysis set (PD) which includes all patients with at least one dose of study drug and evaluable PD data.
Measure: Mean (Standard Deviation); unit: mm^2
Groups:
- LFG316: LFG316 (5 mg/50 µL)
Arm/Group | LFG316 | Sham
Number analyzed (Participants) | 50 | 27
mm^2 | 1.95 (1.01) | 1.58 (1.12)

2. Secondary Outcome: Part A: Change From Baseline in GA Lesions Growth Measured by Fundus Autofluorescence
Description: Mean change in GA lesion growth from baseline to Day 169 and Day 505.
Time Frame: Day 1 to Day 169 and Day 505 (starting from the day of first intravitreal injection until Day 505)
Population: PD Set which included patients who had at least one dose of study drug and had evaluable PD Data.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | LFG316 | Sham
Number analyzed (Participants) | 74 | 38
mm^2
  Day 169 (n=68, 37) | 0.99 (0.60) | 0.88 (0.77)
  Day 505 (n=38, 18) | 2.78 (1.28) | 2.03 (1.00)

3. Secondary Outcome: Part A: Change in Best Corrected Visual Acuity (BCVA) as Measured by the EDTRS (Early Treatment of Diabetic Retinopathy Study) Scale From Baseline to Days 169, 337 & 505 in Patients Receiving Every 28 Days, Successive IVT Doses of LFG316 Compared to Sham
Description: Part A: Summary of best corrected visual acuity over time, statistical analysis of change in best corrected visual acuity over time Parameter: Visual Acuity (EDTRS letter) BCVA scale is 0-100, worst is 0 and best 100 Eye: STUDY
Time Frame: Baseline Day 1, Day 169, Day 337 to Day 505
Population: PD analysis set which includes all patients with at least one dose of study drug and evaluable PD data.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | LFG316 | Sham
Number analyzed (Participants) | 74 | 38
ETDRS letters
  Baseline Day 1 (n=74, 38) | 43.91 (12.93) | 40.26 (14.97)
  Day 169 (n=71, 36) | 48.38 (11.05) | 42.50 (15.14)
  Day 337 (n=53, 30) | 47.49 (11.25) | 42.97 (14.23)
  Day 505 (n=40, 23) | 44.73 (11.29) | 43.78 (14.11)

4. Secondary Outcome: Part A: Summary of Best Corrected Visual Acuity Over Time, Statistical Analysis of Change in Best Corrected Visual Acuity Over Time Parameter: Visual Acuity (EDTRS Letter) BCVA Scale is 0-100, Worst is 0 and Best 100 Eye: FELLOW
Description: Part A: Summary of best corrected visual acuity over time, statistical analysis of change in best corrected visual acuity over time Parameter: Visual Acuity (EDTRS letter) BCVA scale is 0-100, worst is 0 and best 100 Eye: FELLOW
Time Frame: Baseline Day 1, Day 169, Day 337 to Day 505
Population: PD analysis set which includes all patients with at least one dose of study drug and evaluable PD data.
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | LFG316 | Sham
Number analyzed (Participants) | 74 | 38
ETDRS Letters
  Baseline Day 1 (n=74, 38) | 54.66 (22.02) | 55.13 (18.27)
  Day 169 (n=71, 36) | 54.59 (21.92) | 57.33 (17.89)
  Day 337 (n=53, 30) | 52.75 (21.66) | 53.87 (18.83)
  Day 505 (n=40, 23) | 50.95 (20.67) | 49.87 (19.35)

5. Secondary Outcome: Part A: Concentrations of Total LFG316 in Blood During the Course of the Study
Description: Summary statistic of total LFG316 concentrations (pharmacokinetic analysis set)
  n=number of participants, h=hours after the last administered dose e.g.; 0.0 means just before dosing. If the mean concentration is 0.00, that means there is no drug in the bloodstream
Time Frame: Day 1 to Day 559 (starting from the day of first intravitreal injection to day 559)
Population: Pharmacokinetic analysis set: The PK analysis set included all patients with at least one dose of study drug and evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LFG316
Number analyzed (Participants) | 99
ng/mL
  Day 1 (n=99), h=0 | 0.00 (0.00)
  Day 1(n= 97), h= 24 | 293 (332)
  Day 1(n=91), h=336 | 560 (238)
  Day 29 (n=94), h=0 | 289 (214)
  Day 57 (n=96), h=0 | 382 (218)
  Day 85 (n=93), h=0 | 436 (210)
  Day 113 (n=83), h=0 | 433 (219)
  Day 141 (n=84), h=0 | 451 (218)
  Day 141 (n=9), h=672 | 482 (174)
  Day 169 (n=68), h=0 | 446 (204)
  Day 197 (n=73), h=0 | 434 (231)
  Day 225 (n=71), h=0 | 471 (224)
  Day 253 (n=42), h=0 | 465 (237)
  Day 281 (n=69), h=0 | 485 (274)
  Day 309 (n=68), h=0 | 447 (226)
  Day 309 (n=22), h=672 | 405 (189)
  Day 365 (n=40), h=0 | 427 (288)
  Day 393 (n=42), h=0 | 464 (239)
  Day 421(n=40), h=0 | 471 (228)
  Day 449 (n=40), h=0 | 459 (214)
  Day 477 (n=39), h=0 | 422 (236)
  Day 477 (n=41), h=672 | 439 (191)
  Day 477 (n=38), h=1968 | 0.00 (0.00)
  Day 309 (n=16), h=2688 | 0.00 (0.00)
  Day 337 (n=42), h=0 | 435 (283)

6. Secondary Outcome: Part A: Concentrations of Total C5 in Blood During the Course of the Study
Description: Summary statistic of total C5 concentrations n=number of participants, h=scheduled sampling time
Time Frame: Day 1 to Day 559 (starting from the day of first intravitreal injection to day 559)
Population: PD Analysis includes patients who received at least one dose of study drug with evaluable PD data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LFG316 | Sham
Number analyzed (Participants) | 99 | 51
ng/mL
  Day 1 (n=99, 51), h=0 | 147000 (28900) | 142000 (25500)
  (n= 97, 51), h= 24 | 143000 (31200) | 139000 (27600)
  (n=91, 49), h=336 | 149000 (41100) | 136000 (25600)
  Day 29 (n=94, 47), h=0 | 145000 (31200) | 142000 (33900)
  Day 57 (n=96, 49), h=0 | 147000 (29300) | 148000 (40400)
  Day 85 (n=93, 46), h=0 | 154000 (42500) | 144000 (39100)
  Day 113 (n=83, 49), h=0 | 153000 (46200) | 146000 (42100)
  Day 141 (n=84, 45), h=0 | 144000 (32600) | 141000 (25600)
  (n=9, 3), h=672 | 146000 (288000) | 135000 (8000)
  Day 169 (n=68, 37), h=0 | 147000 (39400) | 144000 (38600)
  Day 197 (n=73, 36), h=0 | 143000 (27300) | 139000 (32500)
  Day 225 (n=71, 34), h=0 | 152000 (51600) | 140000 (33600)
  Day 253 (n=42, 18), h=0 | 144000 (38500) | 129000 (31000)
  Day 281 (n=69, 34), h=0 | 145000 (28000) | 144000 (35300)
  Day 309 (n=68, 32), h=0 | 151000 (45200) | 148000 (39400)
  (n=22, 12), h=672 | 137000 (31000) | 145000 (33200)
  Day 365 (n=40, 24), h=0 | 146000 (29300) | 131000 (29300)
  Day 393 (n=42, 22), h=0 | 145000 (23700) | 132000 (28500)
  Day 421(n=40, 22), h=0 | 149000 (24700) | 141000 (34200)
  Day 449 (n=40, 23), h=0 | 160000 (41200) | 144000 (27000)
  Day 477 (n=39, 21), h=0 | 148000 (20400) | 156000 (53900)
  (n=41, 21), h=672 | 158000 (37800) | 155000 (59000)
  (n=38, 22), h=1968 | 198000 (82700) | 186000 (79600)
  Day 309 (n=16, 10), h=2688 | 135000 (19600) | 135000 (18800)
  Day 337 (n=44, 24), h-0 | 147000 (27900) | 137000 (36200)

7. Primary Outcome: Part A: Sensitivity Analysis of the Primary End Point: Mixed Effects Model for Repeated Measurements on GA Lesion Growth Measured by Fundus Autoflourescence
Description: Number is the Estimated Difference (95% CI) in lesion size.
Time Frame: The primary objective was from Day 1 to Day 337, however data was captured to Day 505 as exploratory objective
Population: PD Set which included patients who had at least one dose of study drug and had evaluable PD Data.
Measure: Mean (95% Confidence Interval); unit: mm^2
Groups:
- LFG316 5 Mg-Sham: Difference in mean between LFG316 arm and Sham arm.
Arm/Group | LFG316 | Sham | LFG316 5 Mg-Sham
Number analyzed (Participants) | 50 | 27 | 77
mm^2
  Bilateral Day 169 | 0.975 [.828 to 1.122] | 0.913 [0.712 to 1.114] | 0.062 [-0.184 to 0.308]
  Bilateral Day 337 | 1.825 [1.584 to 2.065] | 1.710 [1.379 to 2.041] | 0.115 [-0.292 to 0.522]
  Bilateral Day 505 | 2.674 [2.314 to 3.034] | 2.506 [2.012 to 3.001] | 0.168 [-0.433 to 0.778]
  Overall Day 169 | 1.036 [0.891 to 1.181] | 0.937 [0.718 to 1.156] | 0.099 [-0.160 to 0.357]
  Overall Day 337 | 1.885 [1.646 to 2.124] | 1.734 [1.397 to 2.070] | 0.152 [-0.259 to 0.562]
  Overall Day 505 | 2.735 [2.376 to 3.094] | 2.530 [2.035 to 3.025] | 0.205 [-0.405 to 0.814]

8. Secondary Outcome: Part B: AUC (Area Under the Curve) - Summary Statistics for PK Parameters
Description: Summary statistic of total LFG316 concentrations (pharmacokinetic analysis set)
  n=number of participants, h=scheduled sampling time
Time Frame: Day 1 to Day 85 (starting from the day of first intravitreal injection to day 85)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- LFG316: LFG316 (10 mg/100 µL)
Arm/Group | LFG316
Number analyzed (Participants) | 7
hr*ng/mL
  AUCall (hr*ng/mL) | 743000 (241000)
  AUClast (hr*ng/mL) | 600000 (212000)

9. Primary Outcome: Part B: Safety and Tolerability of a Single Intravitreal (IVT) Dose of 10 mg/100 μL of LFG316 in Patients With Advanced AMD).
Description: This primary outcome (for Part B) is reported under the Adverse Events section.
Time Frame: Day 1 to Day 85
Measure: Number; unit: number of patients
Groups:
- Part A - LFG316 5mg: Part A - LFG316 5 mg/50 µL injection every 4 weeks for 18 months
- Sham - Part A: sham injection every 4 weeks for a total of 18 injections
- Part B - LFG316 10mg: Part B - LFG316 10 mg/100 µL injection every 4 weeks for 18 months
- Sham - Part B: Single sham injection
Arm/Group | Part A - LFG316 5mg | Sham - Part A | Part B - LFG316 10mg | Sham - Part B
Number analyzed (Participants) | 99 | 51 | 7 | 1
number of patients
  Total # Affected by any Serious Adverse Event | 27 | 11 | 1 | 0
  Total # at Risk by any Serious Adverse Event | 99 | 51 | 7 | 1

10. Secondary Outcome: Tmax (hr)
Description: PART B: Tmax (Time of Maximum concentration observed)
  This is the highest concentration of drug in the blood that is measured after a dose. Cmax usually happens within a few hours after the dose is taken. The time that Cmax happens is referred to as Tmax. For some antiretroviral drugs, a high Cmax is thought to increase the risk of side effects from the drug.
Time Frame: Day 1 to Day 85 (starting from the day of first intravitreal injection to day 85)
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | LFG316
Number analyzed (Participants) | 7
hours | 213 [119 to 311]

11. Secondary Outcome: Part B: Cmax - Summary Statistic for PK Parameters
Description: Summary statistic for Part B of total LFG316 concentrations (pharmacokinetic analysis set) Cmax is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose
Time Frame: Day 1 to Day 85 (starting from the day of first intravitreal injection to day 85)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LFG316
Number analyzed (Participants) | 7
ng/mL | 1010 (213)

12. Secondary Outcome: Part B: Cmax_D - Summary Statistic for PK Parameters
Description: Cmax_D=ng/mL/mg
Time Frame: Day 1 to Day 85 (starting from the day of first intravitreal injection to day 85)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | LFG316
Number analyzed (Participants) | 7
ng/mL/mg | 101 (21.3)

ADVERSE EVENTS:
Groups:
- Part A - Sham: sham injection every 4 weeks for a total of 18 injections
- Part B - LFG316 10mg: Part B - Single LFG316 10 mg/100 µL injection
- Part B - Sham: single sham injection
Arm/Group | Part A - LFG316 5mg | Part A - Sham | Part B - LFG316 10mg | Part B - Sham
Serious Adverse Events (participants affected / at risk) | 27/99 | 11/51 | 1/7 | 0/1
Other Adverse Events (participants affected / at risk) | 98/99 | 42/51 | 4/7 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - LFG316 5mg (N=99) | Part A - Sham (N=51) | Part B - LFG316 10mg (N=7) | Part B - Sham (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Fellow Eye) (Eye disorders) | 1 | 1 | 0 | 0
Visual acuity reduced (Study Eye) (Eye disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Endophthalmitis (Study Eye) (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Auricular haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - LFG316 5mg (N=99) | Part A - Sham (N=51) | Part B - LFG316 10mg (N=7) | Part B - Sham (N=1)
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Macrocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 2 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1 | 0 | 0
Heart valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Corneal dystrophy (Fellow Eye) (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Corneal dystrophy (Study Eye) (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 4 | 2 | 0 | 0
Anterior chamber cell (Study Eye) (Eye disorders) | 3 | 0 | 0 | 0
Anterior chamber flare (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Blepharitis (Fellow Eye) (Eye disorders) | 2 | 0 | 0 | 0
Blepharitis (Study Eye) (Eye disorders) | 4 | 0 | 0 | 0
Blepharitis allergic (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Blepharospasm (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Study Eye) (Eye disorders) | 2 | 1 | 0 | 0
Cataract nuclear (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Cataract nuclear (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Cataract subcapsular (Fellow Eye) (Eye disorders) | 0 | 1 | 0 | 0
Cataract subcapsular (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Charles Bonnet syndrome (Eye disorders) | 1 | 0 | 0 | 0
Charles Bonnet syndrome (Fellow Eye) (Eye disorders) | 0 | 1 | 1 | 0
Charles Bonnet syndrome (Study Eye) (Eye disorders) | 0 | 1 | 1 | 0
Chorioretinal atrophy (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Chorioretinal atrophy (Study Eye) (Eye disorders) | 2 | 1 | 0 | 0
Choroidal neovascularisation (Fellow Eye) (Eye disorders) | 1 | 1 | 0 | 0
Choroidal neovascularisation (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Fellow Eye) (Eye disorders) | 1 | 1 | 0 | 0
Conjunctival haemorrhage (Study Eye) (Eye disorders) | 70 | 29 | 2 | 0
Conjunctival hyperaemia (Study Eye) (Eye disorders) | 3 | 1 | 0 | 0
Conjunctival oedema (Study Eye) (Eye disorders) | 2 | 0 | 0 | 0
Conjunctival vascular disorder (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Corneal deposits (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Corneal oedema (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Corneal opacity (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Corneal scar (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Fellow Eye) (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Study Eye) (Eye disorders) | 1 | 1 | 0 | 0
Dry eye (Fellow Eye) (Eye disorders) | 5 | 2 | 0 | 0
Dry eye (Study Eye) (Eye disorders) | 5 | 3 | 0 | 0
Ectropion (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Erythema of eyelid (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Exfoliation glaucoma (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Eye colour change (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Eye inflammation (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Eye irritation (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Eye irritation (Study Eye) (Eye disorders) | 11 | 5 | 0 | 0
Eye pain (Fellow Eye) (Eye disorders) | 2 | 0 | 0 | 0
Eye pain (Study Eye) (Eye disorders) | 12 | 6 | 0 | 0
Eye pruritus (Fellow Eye) (Eye disorders) | 2 | 1 | 0 | 0
Eye pruritus (Study Eye) (Eye disorders) | 4 | 1 | 0 | 0
Eye swelling (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Eyelid irritation (Study Eye) (Eye disorders) | 2 | 0 | 0 | 0
Eyelid oedema (Study Eye) (Eye disorders) | 2 | 1 | 0 | 0
Eyelids pruritus (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Foreign body sensation in eyes (Study Eye) (Eye disorders) | 10 | 7 | 0 | 0
Glaucoma (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Glaucoma (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Hyphaema (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Iritis (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Keratitis (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Lacrimation decreased (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Lacrimation increased (Study Eye) (Eye disorders) | 6 | 1 | 0 | 0
Macular degeneration (Fellow Eye) (Eye disorders) | 1 | 1 | 0 | 0
Macular oedema (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Neovascular age-related macular degeneration (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Neovascular age-related macular degeneration (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Ocular discomfort (Study Eye) (Eye disorders) | 4 | 2 | 0 | 0
Ocular hyperaemia (Study Eye) (Eye disorders) | 2 | 1 | 0 | 0
Optic disc disorder (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Optic disc haemorrhage (Fellow Eye) (Eye disorders) | 2 | 0 | 0 | 0
Photophobia (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Photophobia (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Photopsia (Study Eye) (Eye disorders) | 1 | 1 | 0 | 0
Posterior capsule opacification (Fellow Eye) (Eye disorders) | 4 | 2 | 0 | 0
Posterior capsule opacification (Study Eye) (Eye disorders) | 3 | 2 | 0 | 0
Pterygium (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Punctate keratitis (Study Eye) (Eye disorders) | 4 | 0 | 0 | 0
Refraction disorder (Fellow Eye) (Eye disorders) | 0 | 1 | 0 | 0
Refraction disorder (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Retinal haemorrhage (Fellow Eye) (Eye disorders) | 2 | 1 | 0 | 0
Retinal haemorrhage (Study Eye) (Eye disorders) | 1 | 0 | 1 | 0
Retinal pigment epitheliopathy (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Retinal pigment epitheliopathy (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Retinal tear (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Scleral hyperaemia (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Subretinal fluid (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Trichiasis (Study Eye) (Eye disorders) | 0 | 1 | 0 | 0
Ulcerative keratitis (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Uveitis (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Study Eye) (Eye disorders) | 1 | 3 | 0 | 1
Visual acuity reduced (Fellow Eye) (Eye disorders) | 3 | 1 | 0 | 0
Visual acuity reduced (Study Eye) (Eye disorders) | 7 | 1 | 0 | 0
Visual acuity reduced transiently (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced transiently (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Visual brightness (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Visual brightness (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment (Study Eye) (Eye disorders) | 3 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 0 | 0
Vitreous detachment (Fellow Eye) (Eye disorders) | 1 | 3 | 0 | 0
Vitreous detachment (Study Eye) (Eye disorders) | 10 | 2 | 0 | 0
Vitreous disorder (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Fellow Eye) (Eye disorders) | 3 | 1 | 0 | 0
Vitreous floaters (Study Eye) (Eye disorders) | 24 | 1 | 1 | 0
Vitreous haemorrhage (Fellow Eye) (Eye disorders) | 1 | 0 | 0 | 0
Vitreous haemorrhage (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Vitreous opacities (Study Eye) (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 3 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tooth deposit (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1 | 0 | 0
Application site pain (Study Eye) (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Fibrosis (Study Eye) (General disorders) | 0 | 1 | 0 | 0
Injection site bruising (Study Eye) (General disorders) | 0 | 1 | 0 | 0
Injection site erythema (Study Eye) (General disorders) | 1 | 0 | 0 | 0
Injection site irritation (Study Eye) (General disorders) | 1 | 0 | 0 | 0
Injection site reaction (Study Eye) (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 6 | 3 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0 | 0
Allergy to chemicals (Immune system disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 4 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 8 | 4 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 0 | 0 | 0
Conjunctivitis (Fellow Eye) (Infections and infestations) | 2 | 0 | 0 | 0
Conjunctivitis (Study Eye) (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 3 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0
Ear infection (Infections and infestations) | 2 | 2 | 0 | 0
Eye infection staphylococcal (Study Eye) (Infections and infestations) | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Hordeolum (Fellow Eye) (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 4 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 13 | 4 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 1
Corneal abrasion (Study Eye) (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 3 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Post procedural complication (Study Eye) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural discomfort (Study Eye) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Study Eye) (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 2 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0 | 0
Intraocular pressure increased (Fellow Eye) (Investigations) | 1 | 0 | 0 | 0
Intraocular pressure increased (Study Eye) (Investigations) | 4 | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Red blood cells urine (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 1 | 0 | 0
Visual acuity tests abnormal (Study Eye) (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Benign neoplasm of eyelid (Fellow Eye) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Eye naevus (Fellow Eye) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 3 | 0 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Visual field defect (Fellow Eye) (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 2 | 0 | 0 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Calculus prostatic (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatic calcification (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Cutis laxa (Fellow Eye) (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Cutis laxa (Study Eye) (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ecchymosis (Study Eye) (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 9 | 3 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Labile hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Poor peripheral circulation (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study conducted in 2 parts, Part A (n=150) & Part B (n=8). Total participants is 158

Primary Outcome for Part B is Safety and Tolerability as presented in the Adverse events section of this report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial